CLINICAL TRIAL: NCT06124391
Title: An Evidence-Based Novel Subtypes of Polycystic Ovary Syndrome and Their Association With Outcomes: a Large Cohort Study
Brief Title: Novel Subtypes of Polycystic Ovary Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Chen Zi-Jiang, Academician, Shandong University
Other Study IDs: PCOS-Subtypes
Record Dates: First submitted 2023-10-26; First posted 2023-11-09 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and plasma samples will be collected.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- HA-PCOS: Patients were classified into each PCOS subtype based on our machine-learning classification model. The feature of the HA-PCOS group is hyperandrogenism.
  Interventions: Other: Long-term follow-up
- OB-PCOS: Patients were classified into each PCOS subtype based on our machine-learning classification model. The feature of the OB-PCOS group is overweight/obesity.
  Interventions: Other: Long-term follow-up
- SHBG-PCOS: Patients were classified into each PCOS subtype based on our machine-learning classification model. The feature of the SHBG-PCOS group is the high level of serum SHBG.
  Interventions: Other: Long-term follow-up
- LH-PCOS: Patients were classified into each PCOS subtype based on our machine-learning classification model. The feature of the LH-PCOS group is the high level of LH and AMH.
  Interventions: Other: Long-term follow-up

INTERVENTIONS:
Other: Long-term follow-up — Participants diagnosed with PCOS were not subjected to any specific intervention post-diagnosis. Instead, they were followed up after 6.5 years to assess various outcomes related to PCOS and associated conditions.

SUMMARY:
To classify subtypes of Polycystic Ovary Syndrome (PCOS) using machine-learning algorithms, and compare the reproductive and metabolic characteristics and IVF outcomes across these identified subtypes.

DETAILED DESCRIPTION:
In this study, we've developed a machine-learning model to classify PCOS patients into four subtypes based on nine clinical characteristics.

The goal of this observational study is to:

* Learn about different PCOS subtypes using our classification model.
* Compare the reproductive and metabolic features of these subtypes.
* Assess the outcomes of IVF among different PCOS subtypes.
* Prospective 6.5-year follow-up data will be collected.

Participants will:

* Undergo a telephone interview to gather details on:

  1. Current physical stats like height and weight.
  2. Reproductive history, including pregnancies and childbirths in recent years.
  3. Details about any IVF treatments.
  4. Current status of conditions such as PCOS, Type 2 Diabetes, hypertension, and dyslipidemia.
* Be invited for a physical examination that includes:

  1. Measurements such as height, weight, blood pressure, and body circumferences.
  2. Laboratory tests for endocrine and metabolic conditions.
  3. Ultrasound scans of the ovaries and liver.

ELIGIBILITY:
Inclusion Criteria:

* PCOS patients diagnosed using the Rotterdam criteria, which requires the presence of at least two of the following:

  1. Menstrual Irregularities: A menstrual cycle length of fewer than 21 days or more than 35 days, and/or fewer than eight cycles per year.
  2. Hyperandrogenism: Defined either by an elevated total testosterone level (as per local laboratory criteria) or by a modified Ferriman-Gallwey (mFG) score of 5 or higher.
  3. Polycystic Ovaries on Ultrasound: Presence of 12 or more follicles measuring 2-9 mm in diameter in each ovary and/or an ovarian volume exceeding 10 mL.

Exclusion Criteria:

Patients with congenital adrenal hyperplasias, androgen-secreting tumours, or Cushing's syndrome) will be excluded.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * Discovery cohort: Patients diagnosed with PCOS who sought care at the Center for Reproductive Medicine, Shandong University between December 2013 and June 2020.
  * The validation cohorts of this study consist of four populations.
    1. China Validation Cohort: Consists of patients from various regions in China, excluding Shandong.
    2. America Validation Cohort: Participants from the Pregnancy in Polycystic Ovary Syndrome II (PPCOS II) trial.
    3. Singapore Validation Cohort.
    4. Europe Validation Cohort: Comprising patients from Turkey.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Persistence of PCOS Diagnosis | At the 6.5-year follow-up visit.
  Determining if patients still meet the Rotterdam criteria for a PCOS diagnosis at the follow-up. The hyperandrogenic, ovulatory, and polycystic ovarian conditions at the follow-up time will be assessed.
Changes in PCOS Subtype | At the 6.5-year follow-up visit.
  Tracking if patients have transitioned between different PCOS subtypes at the follow-up.
Body Mass Index | At the 6.5-year follow-up visit.
  Patients' weight (in kilograms) and height (in meters) will be collected and combined to report BMI in kg/m^2
Non-Alcoholic Fatty Liver Disease (NAFLD) | At the 6.5-year follow-up visit.
  NAFLD will be assessed using abdominal ultrasound.
Hypertension | At the 6.5-year follow-up visit.
  Blood pressure will be assessed, and we will determine if a patient has hypertension, defined as systolic blood pressure (SBP) ≥ 140 mmHg and/or diastolic blood pressure (DBP) ≥ 90 mmHg.
Type 2 Diabetes Mellitus (T2DM) | At the 6.5-year follow-up visit.
  Fasting glucose will be assessed, and we will determine if a patient has T2DM, defined as fasting glucose ≥ 7.0 mmol/l.
Dyslipidemia | At the 6.5-year follow-up visit.
  Defined as the presence of any of the following abnormalities:
  * Total cholesterol ≥ 5.2 mmol/l
  * Triglycerides (TG) ≥ 1.7 mmol/l
  * High-density lipoprotein (HDL) < 1.0 mmol/l
  * Low-density lipoprotein (LDL) ≥ 3.35 mmol/l
Total live birth rate | From the diagnosis of PCOS (at the time of enrollment) until a follow-up period of 6.5 years.
  Live birth is defined as the delivery of any neonate with signs of life at ≥ 28 weeks of gestation.
Clinical pregnancy rate | From the diagnosis of PCOS (at the time of enrollment) until a follow-up period of 6.5 years.
  Clinical pregnancy is defined as the ultrasound confirmation of at least one intrauterine gestational sac.
Pregnancy loss rate | From the diagnosis of PCOS (at the time of enrollment) until a follow-up period of 6.5 years.
  Pregnancy loss is defined as pregnancies that eventuate in a spontaneous abortion or therapeutic abortion that occurred throughout pregnancy.
Maternal and neonatal complications | From the diagnosis of PCOS (at the time of enrollment) until a follow-up period of 6.5 years.
  Any maternal and neonatal complications, including gestational diabetes, preeclampsia, etc., will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Zi-jiang Chen, Study Chair — Center for Reproductive Medicine, Shandong University
Locations (11):
- Penn State College of Medicine, Hershey, Pennsylvania, United States
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Brazil
- China (6):
  - Chengdu Jinjiang Maternity and Child Health Hospital, Chengdu
  - Guangdong Second Provincial General Hospital, Guangzhou
  - Shandong University, Jinan
  - Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai
  - Tianjin Medical University General Hospital, Tianjin
  - General Hospital of Ningxia Medical University, Yinchuan
- National University Hospital, National University of Singapore, Singapore, Singapore
- Karolinska Institutet, Solna, Sweden
- Hacettepe University School of Medicine Hacettepe, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No